CLINICAL TRIAL: NCT04299126
Title: Efficacy and Safety of High Absorption Pad for Blood and Pus With Natural Antimicrobial Agent in Split-thickness Skin Graft Donor Site Wound
Brief Title: Efficacy and Safety of High Absorption Pad in Split-thickness Skin Graft Donor Site Wound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 625/62
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Disorder of Skin Donor Site
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high absorption pad for blood and pus (Experimental): High absorption pad for blood and pus with natural antimicrobial agent composes of sericin and chitosan. It will be covered on half of split-thickness skin graft donor site wound until the wound has healed.
  Interventions: Device: high absorption pad for blood and pus
- commercial wound dressing (Active Comparator): Commercial wound dressing is gauze dressing impregnated with paraffin, containing 0.5% chlorhexidine acetate (Bactigras). It will be covered on half of split-thickness skin graft donor site wound until the wound has healed.
  Interventions: Device: commercial wound dressing

INTERVENTIONS:
Device: high absorption pad for blood and pus — High absorption pad for blood and pus will be covered on half of split-thickness skin graft donor site wound until the wound has healed.
  Arms: high absorption pad for blood and pus
Device: commercial wound dressing — Commercial wound dressing will be covered on half of split-thickness skin graft donor site wound until the wound has healed.
  Arms: commercial wound dressing

SUMMARY:
High absorption pad for blood and pus with natural antimicrobial agent or gauze dressing impregnated with paraffin, containing 0.5% chlorhexidine acetate (Bactigras) will be randomly covered on half of split-thickness skin graft donor site wound. The another will be cover on another half of split-thickness skin graft donor site wound. Then, they will be covered with gauzes and bandage. Time to wound healing, amounts of covered dressing gauzes, signs of infection, pain score, erythema index, melanin index, trans epidermal water loss index, and adverse events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Have split-thickness skin graft donor site wound on thigh
* Age 18-60 years
* Can read and write
* Can follow the study protocol
* Available on appointment date

Exclusion Criteria:

* Systemic infection
* Chronic skin diseases
* Immune deficiency
* Allergic to cellulose, chitosan, sericin, and chlorhexidine
* Psychotic disorders
* Pregnancy or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-03-05 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
wound healing time | not more than 28 days
  The day that the dressing will detach without painful.
amounts of secondary gauze dressing | not more than 28 days
  The amounts of secondary gauze dressing that will be changed because of blood over capacity.

SECONDARY OUTCOMES:
pain score | 5 days after donor site wound was created
  Pain score will be evaluated using visual analogue scale. The 0 and 10 scores mean no pain and very pain, respectively. Higher score means more painful.
signs of infection | not more than 28 days
  Signs of infection mean pain, swollen, red, and warn including pus on the wound.
scar melanin index | 3 months
  Scar melanin index will be measured using Cutometer (Mexameter). There is no unit. Higher value mean higher risk of post inflammatory reaction.
scar erythema index | 3 months
  Scar erythema index will be measured using Cutometer (Mexameter). There is no unit. Higher value mean higher risk of post inflammatory reaction.
transepidermal water loss index | 3 months
  Transepidermal water loss index of scar will be measured using Cutometer (Tewameter). There is no unit. Higher value mean higher risk of unhealthy scar.
scar quality | 3 months
  Scar quality will be evaluated using vancouver scar scale. The 0 and 13 scores mean high scar quality and low scar quality , respectively. Higher score means low scar quality.
adverse events | not more than 28 days
  Adverse events will be observed. They will be recorded as "present" or "not present".
aspartate aminotransferase in serum | not more than 28 days
  Aspartate aminotransferase in serum (in U/L) after treatment will not be more than before treatment.
alanine aminotransferase in serum | not more than 28 days
  Alanine aminotransferase in serum (in U/L) after treatment will not be more than before treatment.
blood urea nitrogen | not more than 28 days
  Blood urea nitrogen (in mg/dl) after treatment will not be more than before treatment.
serum creatinine | not more than 28 days
  Serum creatinine (in mg/dl) after treatment will not be more than before treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No